CLINICAL TRIAL: NCT06785766
Title: Investigating the Effects of Yoga-Based Exercises on Balance, Cognitive Function, Posture, and Body Awareness in Young Adults With Premenstrual Syndrome
Brief Title: Effects of Yoga on Balance, Cognition, Posture, and Body Awareness in Premenstrual Syndrome (PMS)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özlem Çınar Özdemir, Prof.Dr, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yoga for Premenstrual Syndrome
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Premenstrual Syndrome-PMS
Keywords: Quality of life; Premenstrual Syndrome; Yoga; Pain; Cognitive Function; Body Awareness
MeSH Terms: conditions — Premenstrual Syndrome; Pain | interventions — Yoga; Health

STUDY DESIGN:
Intervention Model Description: The women included in the study will be randomized and divided into two groups (arms), 30 participants in each group, as intervention and control groups. Both groups will receive information training at the beginning of the study. The exercise program for the intervention group will consist of 60-minute yoga-based exercise sessions, conducted twice a week for 8 weeks. Additionally, both groups will be instructed to perform a 30-minute walk three times a week.The groups will be formed based on participants' availability, and 8-week yoga flows with gradually increasing difficulty will be applied, based on themes set for each week. Participants assigned to the control group will be asked to continue their routine activities and not to start a new exercise program during the study period. After the second evaluations are completed, the participants in the control group will be offered the opportunity to participate in the yoga program.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The "Intervention Group" will receive an 8-week yoga-based exercise program, consisting of 60-minute sessions held twice a week. Each session includes a 5-minute warm-up, 5 minutes of breathing exercises (pranayama), 40 minutes of yoga postures (asana), 5 minutes of deep relaxation (Savasana), and 5 minutes of meditation. The program will be facilitated by a physiotherapist who will demonstrate the poses, observe participants, and provide verbal instructions for adjustments as needed. The yoga postures will be adapted using props such as blocks, straps, blankets, pillows, and chairs, based on individual needs and abilities. The difficulty of the sessions will gradually increase over the 8 weeks, with the yoga flows being adjusted to match weekly themes and participants' progress.
  Interventions: Behavioral: Yoga-Based Exercise Program
- Control Group (No Intervention): The "Control Group" will not receive any specific intervention during the study period. Participants in this group will be asked to continue their routine activities without starting any new exercise programs. They will be advised to engage in 30-minute walking sessions three times a week as part of their regular routine. No yoga or additional structured exercise will be provided. After the 8-week waiting period, participants in the control group will be given the option to join the yoga-based exercise program if they wish.

INTERVENTIONS:
Behavioral: Yoga-Based Exercise Program — This intervention is an 8-week yoga-based exercise program conducted with 60-minute sessions twice a week. The program aims to improve flexibility, mobility, and overall well-being. Each session consists of 5 minutes of warm-up, 5 minutes of breathing exercises, 40 minutes of yoga postures, 5 minutes of deep relaxation, and 5 minutes of meditation. The intervention adapts yoga postures based on participants' individual needs, offering a flexible approach. The difficulty of the yoga flows gradually increases over the 8 weeks. When necessary, postures are adapted using props like blocks, straps, blankets, and chairs. A physiotherapist guides participants, demonstrating correct techniques and providing verbal instructions. This program combines yoga, breathing exercises, and meditation to enhance physical and mental well-being, promoting long-term health benefits.
  Other Names: 8-Week Yoga Program; Yoga for Health and Wellness; Yoga Therapy for Active Living
  Arms: Intervention Group

SUMMARY:
Premenstrual syndrome (PMS) is characterized by a combination of cognitive, somatic, behavioral, and emotional disorders that occur during the late luteal phase of the menstrual cycle, resolve rapidly after menstruation, and can be severe enough to disrupt daily activities. When reviewing the literature, studies examining the effects of yoga-based exercises on premenstrual syndrome appear to be quite limited. Our aim is to raise awareness among professionals working in this field in our country, contributing to the reduction of symptoms and improvement of the quality of life of individuals with premenstrual syndrome.

DETAILED DESCRIPTION:
Menstruation is a process characterized by symptoms accompanied by emotional, physical, and behavioral changes that occur regularly every month from menarche to menopause, covering an average of 30-35 years of a woman's life. Although menstruation, which constitutes a large period of a woman's life, is a natural physiological cycle, the symptoms that accompany the cycle are among the most common women's health problems.Premenstrual Syndrome (PMS) is defined as 'a condition characterized by distressing physical, behavioral, and psychological symptoms that begin 7-10 days before the menstrual cycle and disappear or significantly decrease with the cessation of menstruation, without being attributed to any underlying psychiatric disorder. Depression, angry outbursts, irritability, anxiety, lack of concentration, and decreased sleep quality are among the most common emotional symptoms of PMS, while physical symptoms include breast tenderness, swelling, fatigue, headache, edema in the extremities, and a feeling of pain or aching. In addition to these frequently seen symptoms in the literature, more than 200 symptoms are defined for PMS. Hormonal fluctuations in women with premenstrual symptoms trigger changes in ligament elasticity, negatively affecting postural balance, coordination and proprioception, and leading to a higher risk of injury. This health issue, which affects many women worldwide, is known to disrupt women's social relationships, increase their tendency to make mistakes or have accidents, reduce work and school performance, and lead to higher rates of sleep problems, substance abuse, criminal behavior, and impaired cognitive functions responsible for memory and emotional control. The etiology of PMS is multifactorial and uncertain, and therefore, there is no definitive treatment method. Although different treatment options are preferred, the aim of the treatment is to relieve the symptoms. Studies have demonstrated that PMS symptoms are more severe in inactive women and that women with severe PMS symptoms are more likely to be inactive. Yoga is one of the oldest methods of personal development, which integrates the body, mind, and spirit, facilitating self-awareness. Yoga increases bodily awareness and cognition as it includes many mind-body exercises such as balancing, stretching, strengthening, physical harmony, breathing and meditation techniques. Studies show that yoga has positive psychological and mental effects on individuals and improves their quality of life. Despite many PMS symptoms negatively impacting a woman's participation in work and social life, there is limited research in the existing literature on specific symptoms. Therefore, this study aims to determine the effectiveness of yoga-based exercises on symptoms in individuals with premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Presence of premenstrual symptoms (scoring 132 or above on the Premenstrual Syndrome Scale (PMSS)),
* Aged 18 and above,
* Able to read and write,
* Willing to participate voluntarily in the study and have signed the informed consent form,
* No problems with cooperation and communication,
* Normal menstrual cycle length (21-35 days) in the past 3 months,
* Not having taken any medications or mineral supplements during the last three menstrual cycles.

Exclusion Criteria:

* Amenorrhea
* Being in the menopausal period
* Pregnancy
* Having given birth
* A diagnosis of cancer
* Having previously practiced yoga
* Having exercise intolerance
* Having received hormone replacement therapy
* Having been enrolled in a physiotherapy program in the past 3 months
* Regular exercise within the past 3 months
* Having musculoskeletal, neurological, serious cardiopulmonary, chronic systemic, psychiatric, balance and coordination, or vestibular system disorders that may prevent participation in exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The Premenstrual Syndrome Scale (PMSS), developed by Gençdoğan (2006) based on DSM-III and DSM-IV-R criteria, is a 44-item, five-point Likert-type scale designed to diagnose PMS and assess symptom severity. Items are rated based on the condition "during the week before menstruation," with responses ranging from 1 - Not at all to 5 - Always.The scale includes nine subdimensions:Depressive affect, anxiety, fatigue, irritability, depressive thoughts, pain, appetite changes, sleep changes, bloating. The total score ranges from 44 to 220, with higher scores indicating more severe symptoms. Scores of 132 or higher (≥50% of the maximum) indicate the presence of PMS.
Body Awareness Questionnaire | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  This questionnaire aims to determine the sensitivity level of body composition, either normal or abnormal, and consists of four subgroups (Changes in body processes, Sleep-wake cycle, Prediction at the onset of illness, Prediction of body responses) with a total of 18 statements. Participants are asked to rate each statement with a score between one and seven. The assessment is scored based on the total points, with higher scores indicating better body sensitivity. The original version of the questionnaire was developed by Shields et al. in 1989. The validity and reliability study for the Turkish version was conducted by Karaca (2017), and the internal consistency coefficient was found to be 0.91.

SECONDARY OUTCOMES:
Demographic Information Form Section C | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The Personal Information Form is a tool created by the researcher to gather data from female participants included in the study, consisting of three sections.
  c) Symptoms Related to PMS
Y Balance Test | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The setup is arranged such that the angle between the anterior and posterior directions is 135˚, and the angle between the posteromedial and posterolateral directions is 90˚. Participants start the test by placing their feet at the center. The individual is instructed to maintain the position of their hands on their hips, keep their feet in contact with the ground, and perform reaches in these three directions while standing on one leg. Traditionally, the test begins with the right foot in the anterior direction, followed by the left foot anterior, right foot posteromedial, left foot posteromedial, right foot posterolateral, and left foot posterolateral directions.Prior to each reach, participants perform 6 practice trials to learn the movement. They are then asked to reach in the anterior, posteromedial, and posterolateral directions three times each. The average reach distance for each direction is calculated, then divided by the leg length and multiplied by 100 to obtain the score.
PostureScreen Mobile Application | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The PostureScreen Mobile application is a validated and reliable tool developed for posture assessment using a camera system on devices with iOS and Android operating systems. The application allows for posture analysis by determining pivot points on photographs taken from the anterior, posterior, and lateral views of the participants. These points are calculated in centimeters and used to display postural deviation values on the phone's screen.
N-Back Test | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The difficulty level in the test is provided by increasing and decreasing the number n. The participant is expected to respond by using the specified buttons when the given stimuli are seen again in a certain order. The N-back test is used to examine working memory processes. Working memory allows information to be temporarily held in the mind with its perceptual, cognitive and emotional aspects and thus to direct behavior. Using the dual n-back task involves remembering a sequence of letters spoken simultaneously and the sequence of positions of a square and determining whether a letter or position matches the one seen before. In addition, optional extended game modes such as Triple N-Back and Arithmetic N-Back can be used for extra difficulty. It also includes features such as statistical tracking, graphics and configurability. The adaptation of the task to Turkish and its transfer to the computer environment were done by Altun and Çevik (2012).
Assessment of Grip Strength | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The Jamar hand dynamometer is recommended by the American Society of Hand Therapists (ASHT) and is considered the gold standard due to its high reliability. According to the procedure, the participant will be seated on a chair without a backrest, with the arm to be evaluated positioned in adduction close to the body, the elbow flexed at 90°, and the forearm and hand in mid-rotation. The participant's hand will be placed on the dynamometer, and they will be instructed to squeeze the dynamometer with full force for three seconds without holding their breath. During this time, the evaluator will provide standard verbal cues such as "Stronger!" and "Continue!" At the end of three repetitions, the highest result will be accepted as the maximum grip strength. A 15-second rest period will be given between each trial to prevent muscle fatigue, and the grip strength will be recorded in kilograms on the data recording form.
Stabilizer Pressure Biofeedback Unit | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The 5-level core stabilization test developed by Sahrmann is used to assess participants' core stability levels. Participants will be trained to follow the standard protocol by Aggarwal et al. In this study, they will start in a supine hook-lying position with the stabilizer aligned to the natural lordotic curve and inflated to 40 mmHg. After learning abdominal curling, participants must maintain abdominal pressure within a 10 mmHg deviation. To advance to the next level, pressure must not exceed a 10 mmHg deviation from 40 mmHg. If the deviation exceeds 10 mmHg, the test will end. Three attempts will be made per level, with a 1-minute rest between transitions to account for fatigue.
Cough Strength | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  Cough strength will be assessed using a peak cough flow meter (PEF meter) (ExpiRite Peak Flow Meter, China) while participants are seated in a supported chair. Participants will first be instructed and shown how to cough as forcefully as possible into the PEF meter after taking a deep breath. The peak flow rate (PEF) achieved during the coughing maneuver will then be recorded. The test will be repeated at least three times, and the highest value will be recorded for analysis. A disposable mouthpiece will be used for each participant, and a 30-second rest period will be provided between measurements to prevent participant fatigue. The peak cough flow meter measures values between 60 and 800 L/min. The normal value for adults is >360 L/min. Values <270 L/min are considered indicative of ineffective coughing, and the use of cough assistive devices is recommended. If the measurement is <160 L/min, airway clearance is considered not to have occurred .
Joint Position Sense Test | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The joint position sense measurement will be conducted using a digital goniometer, targeting hip joint angles of 30°, 45°, and 60°. The test will take place in a controlled, quiet environment with participants positioned in the supine posture. To eliminate visual cues of leg movements, participants' eyes will be covered with a black band during the measurement process. When the participant's knee is in extension, the rotation center of the goniometer will be positioned at the rotation center of the knee joint. The target angle for each measurement will be stated before the test, and the specific angle will be demonstrated to the participant twice before each measurement. Following this, the participant will be asked to replicate the target angles three times, and the deviation from the target angle will be recorded for all angle values. Measurements will be taken for both lower extremities.
Premenstrual Symptoms Impact Survey (PMSIS) | The scale will be administered at baseline (prior to the start of the 8-week yoga program) and after the completion of the program (week 8).
  The Premenstrual Symptoms Impact Survey (PMSIS) was developed by Wallenstein et al. in 2008 to assess the impact of premenstrual symptoms on quality of life. It consists of six questions and uses a five-point Likert scale. The total score obtained from the scale ranges from 6 to 30, which is then converted to a score between 0 and 100. Higher scores indicate a worsening of quality of life. The validity and reliability study of the scale was conducted by Güler et al. in 2015. The Cronbach's alpha value for the scale, as determined by Güler et al., is 0.89.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem ÇİNAR ÖZDEMİR, Prof. Dr., PhD, Study Director — İzmir Democracy University
Locations (1):
- Siirt University, Siirt, Si̇i̇rt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hopkins BB, Vehrs PR, Fellingham GW, George JD, Hager R, Ridge ST. Validity and Reliability of Standing Posture Measurements Using a Mobile Application. J Manipulative Physiol Ther. 2019 Feb;42(2):132-140. doi: 10.1016/j.jmpt.2019.02.003. Epub 2019 Apr 15. PMID 31000345
- [Background] Colucci DB, Fiore JF Jr, Paisani DM, Risso TT, Colucci M, Chiavegato LD, Faresin SM. Cough impairment and risk of postoperative pulmonary complications after open upper abdominal surgery. Respir Care. 2015 May;60(5):673-8. doi: 10.4187/respcare.03600. Epub 2015 Feb 10. PMID 25669217
- [Background] Aoki M, Suzuki M, Suzuki S, Takao H, Okayama H. Cognitive function evaluation in premenstrual syndrome during the follicular and luteal phases using near-infrared spectroscopy. Compr Psychoneuroendocrinol. 2022 Feb 4;10:100117. doi: 10.1016/j.cpnec.2022.100117. eCollection 2022 May. PMID 35755198
- [Background] Friden C, Hirschberg AL, Saartok T, Backstrom T, Leanderson J, Renstrom P. The influence of premenstrual symptoms on postural balance and kinesthesia during the menstrual cycle. Gynecol Endocrinol. 2003 Dec;17(6):433-9. doi: 10.1080/09513590312331290358. PMID 14992161
- [Background] Kroll-Desrosiers AR, Ronnenberg AG, Zagarins SE, Houghton SC, Takashima-Uebelhoer BB, Bertone-Johnson ER. Recreational Physical Activity and Premenstrual Syndrome in Young Adult Women: A Cross-Sectional Study. PLoS One. 2017 Jan 12;12(1):e0169728. doi: 10.1371/journal.pone.0169728. eCollection 2017. PMID 28081191